CLINICAL TRIAL: NCT02116413
Title: Does the Time Between the End of Vascular Filling and Evaluation of Its Effectiveness Modify Fluid Challenge Results in Septic Shock?
Acronym: FC-Rev
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/CR-01; 2013-A01702-43 (Other: ANSM)
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2016-01

CONDITIONS: Septic Shock
Keywords: fluid challenge; fluid resuscitation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population consists of patients admitted to intensive care, sedated and under controlled ventilatory support with septic shock criteria defined by severe sepsis associated with hypotension despite fluid resuscitation of 20-40 ml / kg and requiring vascular filling according to the following criteria:
  oliguria <0.5 ml / kg / h for at least 2h skin mottling Arterial Lactate > 2 mmol / l SvcO2 <70% or SvO2 <65% Patient on noradrenaline.
  Severe sepsis is defined as a systemic inflammatory response associated with a suspected or proven infection and hypotension before filling, a lactate> 4 mmol / l or organ dysfunction.
  Intervention: Fluid challenge Intervention: Cardiac ultrasound
  Interventions: Procedure: Fluid challenge; Procedure: Cardiac ultrasound

INTERVENTIONS:
Procedure: Fluid challenge — The fluid challenge starts at minute 0 (T0) and consists of 500ml of crystalloids over 10 minutes.
Procedure: Cardiac ultrasound — Ultrasound measures are made at T0, T2, T4, T6, T8, T10, T20 and T30.

SUMMARY:
The main objective of this study is to evaluate in a population of patients with septic shock receiving 500 ml crystalloid over 10 minutes, the proportion of patients classified as "responders" to the fluid challenge (increase of at least 15% of ITV in aortic) at the end of vascular filling (T10) and becoming "non-responders" 20 minutes after the end of the fluid challenge (T30) and whether this proportion is greater than 10 points.

DETAILED DESCRIPTION:
The secondary objectives of this study are :

A. To assess changes in different ultrasound parameters: E wave , E / A ratio , E / E ' in the event of vascular filling and construct a dose response curve for vascular filling.

B. To determing a threshold value for the mitral E wave velcoity that can predict a positive response to volume expansion at T10 defined by a 15% increase in the sub aortic velocity time integral (ITV) after 500 ml of crystalloids in 10 minutes.

C. To determine a threshold value for theITV at T0 that can predict a positive response to volume expansion at T10 defined by a 15% increase in the ITV after 500 ml of crystalloids in 10 minutes.

D. To evaluate the proportion of responders at T10 becoming non-responders at T20.

E. To evaluate the proportion of nonresponders at T10 and responders at T30 .

F. To estimate the proportion of patients changing status regardless of the direction of change between T10 and T30 .

ELIGIBILITY:
Inclusion Criteria:

* The patient has given his/hers consent or the patient is in an emergency situation (commitment to obtain the consent of the patient as soon as his/her condition permits)
* Patient affiliated or beneficiary of a health insurance plan
* Patient with septic shock: proven or suspected infection associated with hypotension or lactate> 4 mmol / l or organ dysfunction. Hypotension despite fluid resuscitation of 20 to -40 ml / kg.
* Patient under controlled mechanical ventilation
* Patient requiring vascular filling according to the following criteria:
* oliguria <0.5 ml / kg / h for at least 2h
* skin mottling
* Arterial Lactate > 2 mmol / l
* SvcO2 <70% or SvO2 <65%
* Patient on noradrenaline.

Exclusion Criteria:

* The patient is has in another interventional study that might change the results of this study within the past 3 months
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* The patient is pregnant, parturient, or breastfeeding
* Valvular pathology: grade III and IV aortic or mitral insufficiency
* Non sinus electrocardiogram
* Non-echogenic patient
* Patient with any spontaneous breathing
* Moribund patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients admitted to intensive care, sedated and under controlled ventilatory support with septic shock criteria defined by severe sepsis associated with hypotension despite fluid resuscitation of 20-40 ml / kg and requiring vascular filling according to the following criteria:
  * oliguria <0.5 ml / kg / h for at least 2h
  * skin mottling
  * Arterial Lactate > 2 mmol / l
  * SvcO2 <70% or SvO2 <65%
  * Patient on noradrenaline.
  Severe sepsis is defined as a systemic inflammatory response associated with a suspected or proven infection and hypotension before filling, a lactate> 4 mmol / l or organ dysfunction.
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01-08 (Actual); Study Completion 2016-01-08 (Actual)

PRIMARY OUTCOMES:
Patient status changes from "responder" at the end of the fluid challenge (T10) to "non-responder" 20 minutes after the end of the fluid challenge (T30). | 30 minutes

SECONDARY OUTCOMES:
Mitral E wave | Baseline (minute 0)
Mitral E wave | 2 minutes
Mitral E wave | 4 minutes
Mitral E wave | 6 minutes
Mitral E wave | 8 minutes
Mitral E wave | 10 minutes
Mitral E wave | 20 minutes
Mitral E wave | 30 minutes
Mitral A wave | Baseline (minute 0)
Mitral A wave | 2 minutes
Mitral A wave | 4 minutes
Mitral A wave | 6 minutes
Mitral A wave | 8 minutes
Mitral A wave | 10 minutes
Mitral A wave | 20 minutes
Mitral A wave | 30 minutes
E' Wave at the lateral mitral annulus | Baseline (minute 0)
E' Wave at the lateral mitral annulus | 2 minutes
E' Wave at the lateral mitral annulus | 4 minutes
E' Wave at the lateral mitral annulus | 6 minutes
E' Wave at the lateral mitral annulus | 8 minutes
E' Wave at the lateral mitral annulus | 10 minutes
E' Wave at the lateral mitral annulus | 20 minutes
E' Wave at the lateral mitral annulus | 30 minutes
ITV | Baseline (minute 0)
ITV | 10 minutes
ITV | 20 minutes
ITV | 30 minutes
Patient status changes from "responder" at the end of the fluid challenge (T10) to "non-responder" 10 minutes after the end of the fluid challenge (T20). | 20 minutes
Patient status changes from "non-responder" at the end of the fluid challenge (T10) to "responder" 20 minutes after the end of the fluid challenge (T30). | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (9):
- France (9):
  - CHU d'Amiens - Hôpital Nord, Amiens
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - CHU de Clermont Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - APHM - Hôpital Nord, Marseille
  - CHU de Nantes - Hôpital Guillaume et René Laennec, Nantes
  - CHU de Nice - Hôpital St-Roch, Nice
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Roger C, Zieleskiewicz L, Demattei C, Lakhal K, Piton G, Louart B, Constantin JM, Chabanne R, Faure JS, Mahjoub Y, Desmeulles I, Quintard H, Lefrant JY, Muller L; AzuRea Group. Time course of fluid responsiveness in sepsis: the fluid challenge revisiting (FCREV) study. Crit Care. 2019 May 16;23(1):179. doi: 10.1186/s13054-019-2448-z. PMID 31097012